CLINICAL TRIAL: NCT00660647
Title: Optimized Treatment Algorithm in Early Rheumatoid Arthritis: Methotrexate and Intra-articular Glucocorticosteroid Plus Adalimumab or Placebo in the Treatment of Early Rheumatoid Arthritis
Brief Title: Optimized Treatment Algorithm for Patients With Early Rheumatoid Arthritis (RA)
Acronym: OPERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Abbott (Industry); Meda Pharmaceuticals (Industry); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VEK-20070008
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis, adalimumab, efficacy, adverse events
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methotrexate + adalimumab (Experimental): Methotrexate and intraarticular triamcinolone hexacetonide plus adalimumab.
  Interventions: Drug: Adalimumab
- methotrexate + placebo (Placebo Comparator): Methotrexate and intraarticular triamcinolone hexacetonide and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — Adalimumab injection 0.8 ml (40 mg) s.c. every second week in up to 2 years
  Other Names: Humira
  Arms: methotrexate + adalimumab
Drug: Placebo — Saline injection 0.9%, 0.8 ml s.c. every second week up to 2 years
  Other Names: Saline
  Arms: methotrexate + placebo

SUMMARY:
Optimized treatment algorithm in early rheumatoid arthritis:

Methotrexate and intra-articular glucocorticosteroid plus adalimumab or placebo in the treatment of early rheumatoid arthritis.

A Randomised, double-blind and placebo-controlled, two arms, parallel group study of the additive effect of adalimumab concerning inflammatory control and inhibition of erosive development.

Optimized Treatment Algorithms for Patients with Early RA

DETAILED DESCRIPTION:
In newly diagnosed rheumatoid arthritis patients it is recommended to treat as soon as possible with methotrexate and steroids However, this treatment algorithm, will only bring one third of the patients into remission and cannot stop progressive, persistent joint damage. The possible benefits and risks of adding adalimumab to this conventional treatment algorithm is unknown.

The aim of the study is to clarify the possible benefits of adding adalimumab an anti-TNF-alfa inhibitor versus placebo to the treatment of rheumatoid arthritis patients, who are treated very early and given methotrexate and intraarticular triamcinolone hexacetonide. Efficacy will be evaluated by DAS 28, ACR 20/50/70, HAQ, progressive changes in X-ray, MRI and DXA-scans.

Adverse events will also be registered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (more than 18 years) with rheumatoid arthritis according to the ACR classification criteria (1) who have had the diagnose < 6 months.

2. Moderate to severe rheumatoid arthritis defined as DAS28 (CRP-based) > 3.2.

3. Negative pregnancy test (serum HCG) for women of childbearing potential prior to trial start. (Non-fertile women are defined as postmenopausal for at least 1 year or surgical sterilisation (bilateral tubal ligation, bilateral oophorectomy or hysterectomy)). Fertile women included in the trial should use contraception during the entire trial period (i.e. one of the following methods: Oral contraception, intrauterine device (IUD), depot injection of progesterone, subdermal implantation, contraceptive vaginal ring, transdermal depot plaster). In addition, contraception should be used for a period of 150 days after any discontinuation of trial medicine.

4. Ability and willingness to inject the sc. injections him/herself or to have an assistant give the injections.

5. Ability and willingness to give written informed consent and to meet the requirements of the trial protocol.

Exclusion Criteria:

1. Persons with latent TB defined with a positive Mantoux test (>12 mm for vaccinated and 6 mm for non-vaccinated), positive cultivation of mycobacteria in tissue samples, chest X-ray indicating TB,or other risk factors for activation of untreated latent TB, and persons not been given adequate TB prophylaxis according to the instructions of the department.

2. Active or recurrent infections or severe infections requiring hospitalization or treatment with i.v. antibiotics within the last 30 days or oral antibiotics within the last 14 days prior to inclusion

3. Positive serology for Hepatitis B or C indicating active infection.

4. Medical history with a positive HIV status (Check of HIV test upon suspicion).

5. Medical history with histoplasmosis or listeriosis.

6. Previous cancer or lymph proliferative disease except cases teated radically and have been without relapse for a minimum of 5 years.

Patients with previous squamous cell carcinoma, basal cell skin carcinoma or cervical dysplasia, who have been treated successfully and radically can be included.

7. Previous diagnosis or signs of demyelinized disease in the CNS system (e.g. optic neuritis, visual disorder, disturbed gait, facial paralysis, apraxia).

8. Severe renal insufficiency (creatinine clearance < 35 ml/min - nomogram).

9. Affected liver function: Liver enzymes > 2 x above normal limit value.

10. Clinical significant drug or alcohol abuse during the past year and/or current daily alcohol consumption.

11. Unstable diabetes, unstable ischemic heart disease, heart insufficiency (NYHA III-IV), active chronic inflammatory intestinal disease, recent cerebral apoplexia (within 3 months), chronic leg ulcer or any other condition (e.g. kateter a demeure)which according to the investigator imposes an increased risk to the subject, if he/she participates in the protocol.

12. Anticoagulant therapy.

13. Pregnancy or breast-feeding.

14. Other inflammatory rheumatic diseases.

15. Aggressive parvovirus B19 infection.

16. Previous treatment with one or more DMARDs.

17. Glucocorticosteroid treatment within the last 4 weeks (except nasal and inhalation steroids).

18. Contraindications for trial medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve a DAS28 < 3.2 | 0, 1, 3, 6, 9, 12 and 24 months (DAS28)

SECONDARY OUTCOMES:
Changes in DAS28 from start of treatment | 1, 3, 6, 9, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Stengaard-Pedersen, Professor, Principal Investigator — Aarhus University/Aarhus University Hospital; Kim Hørslev-Petersen, Professor, Principal Investigator — King Christian X's Rheumatism Hospital, Graasten, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Skejoe C, Hansen AS, Stengaard-Pedersen K, Junker P, Hoerslev-Pedersen K, Hetland ML, Oestergaard M, Greisen S, Hvid M, Deleuran M, Deleuran B. T-cell immunoglobulin and mucin domain 3 is upregulated in rheumatoid arthritis, but insufficient in controlling inflammation. Am J Clin Exp Immunol. 2022 Jun 15;11(3):34-44. eCollection 2022. PMID 35874466
- [Derived] Masic D, Stengaard-Pedersen K, Logstrup BB, Horslev-Petersen K, Hetland ML, Junker P, Ostergaard M, Ammitzboll C, Moller S, Christensen R, Ellingsen T. Similar lipid level changes in early rheumatoid arthritis patients following 1-year treat-to-target strategy with adalimumab plus methotrexate versus placebo plus methotrexate: secondary analyses from the randomised controlled OPERA trial. Rheumatol Int. 2021 Mar;41(3):543-549. doi: 10.1007/s00296-020-04756-5. Epub 2021 Jan 2. PMID 33386898
- [Derived] Sode J, Krintel SB, Carlsen AL, Hetland ML, Johansen JS, Horslev-Petersen K, Stengaard-Pedersen K, Ellingsen T, Burton M, Junker P, Ostergaard M, Heegaard NHH. Plasma MicroRNA Profiles in Patients with Early Rheumatoid Arthritis Responding to Adalimumab plus Methotrexate vs Methotrexate Alone: A Placebo-controlled Clinical Trial. J Rheumatol. 2018 Jan;45(1):53-61. doi: 10.3899/jrheum.170266. Epub 2017 Nov 15. PMID 29142030
- [Derived] Glinatsi D, Baker JF, Hetland ML, Horslev-Petersen K, Ejbjerg BJ, Stengaard-Pedersen K, Junker P, Ellingsen T, Lindegaard HM, Hansen I, Lottenburger T, Moller JM, Ornbjerg L, Vestergaard A, Jurik AG, Thomsen HS, Torfing T, Moller-Bisgaard S, Axelsen MB, Ostergaard M. Magnetic resonance imaging assessed inflammation in the wrist is associated with patient-reported physical impairment, global assessment of disease activity and pain in early rheumatoid arthritis: longitudinal results from two randomised controlled trials. Ann Rheum Dis. 2017 Oct;76(10):1707-1715. doi: 10.1136/annrheumdis-2017-211315. Epub 2017 Jun 13. PMID 28611080
- [Derived] Horslev-Petersen K, Hetland ML, Ornbjerg LM, Junker P, Podenphant J, Ellingsen T, Ahlquist P, Lindegaard H, Linauskas A, Schlemmer A, Dam MY, Hansen I, Lottenburger T, Ammitzboll CG, Jorgensen A, Krintel SB, Raun J, Johansen JS, Ostergaard M, Stengaard-Pedersen K; OPERA Study-Group. Clinical and radiographic outcome of a treat-to-target strategy using methotrexate and intra-articular glucocorticoids with or without adalimumab induction: a 2-year investigator-initiated, double-blinded, randomised, controlled trial (OPERA). Ann Rheum Dis. 2016 Sep;75(9):1645-53. doi: 10.1136/annrheumdis-2015-208166. Epub 2015 Oct 21. PMID 26489704
- [Derived] Ammitzboll CG, Steffensen R, Bogsted M, Horslev-Petersen K, Hetland ML, Junker P, Johansen JS, Podenphant J, Ostergaard M, Ellingsen T, Stengaard-Pedersen K. CRP genotype and haplotype associations with serum C-reactive protein level and DAS28 in untreated early rheumatoid arthritis patients. Arthritis Res Ther. 2014 Oct 31;16(5):475. doi: 10.1186/s13075-014-0475-3. PMID 25359432
- [Derived] Laustsen JK, Rasmussen TK, Stengaard-Pedersen K, Horslev-Petersen K, Hetland ML, Ostergaard M, Junker P, Hvid M, Deleuran B. Soluble OX40L is associated with presence of autoantibodies in early rheumatoid arthritis. Arthritis Res Ther. 2014 Oct 30;16(5):474. doi: 10.1186/s13075-014-0474-4. PMID 25359291
- [Derived] Greisen SR, Schelde KK, Rasmussen TK, Kragstrup TW, Stengaard-Pedersen K, Hetland ML, Horslev-Petersen K, Junker P, Ostergaard M, Deleuran B, Hvid M. CXCL13 predicts disease activity in early rheumatoid arthritis and could be an indicator of the therapeutic 'window of opportunity'. Arthritis Res Ther. 2014 Sep 24;16(5):434. doi: 10.1186/s13075-014-0434-z. PMID 25249397
- [Derived] Ammitzboll CG, Thiel S, Jensenius JC, Ellingsen T, Horslev-Petersen K, Hetland ML, Junker P, Krogh NS, Ostergaard M, Stengaard-Pedersen K. M-ficolin levels reflect disease activity and predict remission in early rheumatoid arthritis. Arthritis Rheum. 2013 Dec;65(12):3045-50. doi: 10.1002/art.38179. PMID 24022747